CLINICAL TRIAL: NCT05960643
Title: Health Belief Model on Breast Examination Skills
Brief Title: The Effect of Education Given According to the Health Belief Model on Breast Examination Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahide Akeren (Other)
Responsible Party: Sponsor-Investigator, Zahide Akeren, Lecturer Doctor, Bayburt University
Organization: Bayburt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BREAST EXAMINATION SKILLS; Bayburt University (Other: Bayburt University)
Record Dates: First submitted 2023-06-15; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Self-Examination
Keywords: breast examination; Health Belief Model; skill
MeSH Terms: conditions — Breast Self-Examination

STUDY DESIGN:
Intervention Model Description: The sample size of the study was calculated in the G*Power 3.1.9.7 program such that the error amount was α=0.05, the power of the test was 0.80 (80%) and the effect size was 0.60. As a result of the statistical analysis, it was found that a total of 90 students, 45 in the experimental group and 45 in the control group, should be included in the study. Considering that if the sample size increases, the standard error will decrease and the working power will increase, each group was increased by 22% (10 people) and it was planned to include 110 students in the study, 55 students for each group. In the first stage, the sample consisted of 148 students who agreed to participate in the study. In the second phase of the study, the sample was planned to consist of 110 female students selected by simple and stratified randomization method (55 experimental, 55 control).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast self-examination group (Experimental): This group was planned to consist of 51 female students studying at the university. First of all, students will be contacted through their electronically registered contact information. In the pre-test, the researchers will apply the 'Personal Information Form' and the 'Health Belief Model Scale' to the students with the self-report method. Afterwards, students will be given BSE training consisting of two 120-minute sessions. In the first session of the training, theoretical trainings about breast cancer and BSE will be given for 30 minutes. In the second session, BSE application will be shown on the wearable breast model and each student will practice on the model. The practice skills of the participants will be evaluated by the researchers using the 'BSE Practice Skill Evaluation Form'. At the end of the 'Health Belief Model Scale' application, face-to-face and 3 weeks later, online applications will be filled as a post-test.
  Interventions: Other: Training and application in breast modeling
- Control group (Active Comparator): No intervention will be made against people in this group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Training and application in breast modeling — BSE application skill evaluation form will be evaluated out of 100 points. The form includes 7 skills: carefully reviewing the model, using three types of pressure, massage, hand position, performing three types of movement, examining each breast for five minutes, and detecting the nodule in the model. A high score is interpreted as a high level of skills.
  Other Names: Experimental: Breast self-examination group
  Arms: Breast self-examination group
Other: Control — No intervention will be made against people in this group.
  Arms: Control group

SUMMARY:
The randomized controlled study to examine the effects of the educational interventions on BSE by revealing the breast self-examination (BSE) practices and breast health beliefs of female students studying at the university were completed with 101 students, 51 of whom were in the "experimental" and 50 "control" groups. The data were collected between November and December 2022 at a university in the Eastern Black Sea region of Turkey, using the 'Personal Information Form', 'BSE Practice Skill Assessment Form' and the 'Health Belief Model Scale' as a pre-test. As an initiative, 'BSE training given according to the Health Belief Model', which includes 120 minutes of training, including theoretical and model-based BSE practice, was implemented. Then, 3 weeks later, the 'BSE Application Skill Evaluation Form' was applied as a post-test. Data were analyzed using Indepent Sample and Paired Sample t-test, Benferroni test, Pearson correlation analysis.

DETAILED DESCRIPTION:
Materials and Methods Type of Research The research was carried out in a randomized controlled manner in order to reveal the breast self-examination (BSE) practices and breast health beliefs of female university students and to examine the effects of educational interventions on BSE.

Place and Time of Research The data of the research were collected at a university located in the Eastern Black Sea region of Turkey between December 2022 and January 2023.

Population and Sample of the Research The universe of the research consisted of female students studying at a university located in the Eastern Black Sea region of Turkey. The number of samples was calculated in the G*Power 3.1.9.7 program so that the error amount was α=0.05, the power of the test was 0.80 (80%) and the effect size was 0.60. As a result of the statistical analysis, it was found that a total of 90 students, 45 in the experimental group and 45 in the control group, should be included in the study. Considering that if the sample size increases, the standard error will decrease and the working power will increase, each group was increased by 22% (10 people) and a total of 110 students, 55 students for each group, were included in the study. The 'simple and stratified sampling' method was used as the randomization method. Simple and stratified randomization method was used in the planning of the research sample. Experimental and control groups within the scope of the study were determined by simple randomization method (coin-toss). In the first stage, the sample consisted of 148 students who agreed to participate in the study. In the second phase of the study, the sample consisted of 110 female students (55 experimental, 55 control) who were selected by simple and stratified randomization method and who had not received BSE training and breast cancer diagnosis according to the Health Belief Model.

Data Collection Tools The data were collected using the 'Personal Information Form' and the 'Health Belief Model Scale', and the 'BSE Practice Skills Evaluation Form' for the students in the experimental group. As an initiative, 'BSE training given according to the Health Belief Model' was carried out.

Personal Information Form This form was created by researchers by scanning the literature. There are 5 questions in the form: age, class, marital status, age at first menstruation, presence of breast cancer diagnosis in the family.

BSE Practice Skill Evaluation Form This form, which was created by the researchers by scanning the literature as a guide to the application made by the students on the wearable breast model, was evaluated over 100 points. The form included 7 skills: carefully reviewing the model, using three types of pressure, massage, hand position, performing three types of movement, examining each breast for five minutes, and detecting the nodule in the model. The high score was interpreted as having high skills.

Health Belief Model Scale (HBMS) This scale was first developed by Champion in 1984 based on the Health Belief Model. The scale has 8 dimensions: sensitivity, caring, health motivation, BSE barriers, benefits, self-efficacy, mammography benefits and barriers.

Breast Self Examination Training The training included 120 minutes of training on normal breast, breast cancer risk factors, symptoms, etiology, treatment, the role of healthy lifestyles in preventing breast cancer, screening and early diagnosis methods, BSE methods and BSE on a model.

Data Collection Method Experimental Group Data Collection Method This group consisted of 51 female students studying at a university located in the Eastern Black Sea region of Turkey. First of all, students were reached from their electronically registered contact information. On the day of the start of the training, the 'Personal Information Form' and the 'Health Belief Model Scale' as a pre-test were administered to the students by face-to-face interview method by the researchers. Afterwards, the students were given BSE training consisting of two 120-minute sessions. In the first session of the training, theoretical trainings on breast cancer and BSE were given for 30 minutes. In the second session, BSE application was shown on the wearable breast model and each student practiced on the model. The application was evaluated using the 'BSE Application Skill Evaluation Form'. At the end of the "Health Belief Model Scale" application, face-to-face and 3 weeks later, online applications were filled as a post-test.

Control Group Data Collection Method This group consisted of 50 female students studying at a university located in the Eastern Black Sea region of Turkey. First of all, students were reached from their electronically registered contact information. The 'Personal Information Form' and the 'Health Belief Model Scale' as a pre-test were filled in by online applications by the researchers. The individuals in this group did not receive any intervention. As a post-test, the Health Belief Model Scale was filled in online applications 3 weeks later as a post-test.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in the study are that female students studying at a university in the Eastern Black Sea region of Turkey continue their education and have their contact addresses, have not received BSE training according to the Health Belief Model, have not been diagnosed with breast cancer, and agree to participate in the research.

Exclusion Criteria:

* Students were excluded from the study if they did not want to continue the research at any stage of the study and were diagnosed with breast cancer.

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Breast Self Examination Practice Skill
Enrollment: 101 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Breast Self Examination Practice Skill Assessment | Three weeks
  The form was created by the researchers by scanning the literature as a guide to the application made by the students on the wearable breast model. The form will be evaluated out of 100 points. The form includes 7 skills: carefully reviewing the model, using three types of pressure, massage, hand position, performing three types of movement, examining each breast for five minutes, and detecting the nodule in the model. A high score is interpreted as a high level of skills.

SECONDARY OUTCOMES:
Health Belief Model Scale | Three weeks
  The scale does not have a grand total score. Each dimension uses its own total score. Sensitivity, caring, health motivation, BSE benefits, BSE barriers and BSE self-efficac were used. The scale is 5-point Likert type. A score closer to 5 means that sensitivity, caring, health motivation, BSE benefits, BSE barriers and BSE self-efficacy are perceived to be high.

CONTACTS AND LOCATIONS:
Overall Officials: Bayburt University, Study Chair — Bayburt University
Locations (1):
- Bayburt University, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov/18928520/